CLINICAL TRIAL: NCT05653934
Title: Virtual Reality Immersion With 360° Virtual Reality Headset to Reduce Postoperative Anxiety and Pain After Surgery for Colorectal Cancer: a Randomized Controlled Pilot Trial - VIREA Trial
Brief Title: Use of VIrtual REAlity to Reduce Postoperative Anxiety and Pain After Surgery for Colorectal Cancer
Acronym: VIREA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: VR 4 GOOD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP211134; IDRCB 2021-A01436-35 (Registry Identifier: ANSM)
Record Dates: First submitted 2022-10-03; First posted 2022-12-16 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Colon Tumor, Malignant; Rectum Tumor; Pain, Postoperative
Keywords: colon cancer; anxiety; pain; virtual reality; malignant colon tumor; malignant rectum tumor; virtual reality immersion
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Pain, Postoperative; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Determine if virutal reality help reduce postoperative anxiety in patients operated for colorectal cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive reality group (Experimental): patients receive care according to the usual practices of the department as well as virtual reality. Virtual reality immersion offers a visual and auditory experience during a soothing journey through visual worlds filmed in natural environments. Virtual reality headset is put on the day before the operation and in the morning just before going to the operating theatre (only on the morning of the operation for patients hospitalized the same day). The colorectal cancer surgery then proceeds as usual. In the postoperative period, virtual reality sessions are offered every day and on request without any limit in number (day and night).
  Interventions: Behavioral: Pre-operative use of virtual reality headset; Procedure: Standard surgery; Behavioral: Post-operative use of virtual reality headset
- Standard care group (Active Comparator): patients are treated according to usual practices of the department and do not have access to virtual reality.
  Interventions: Procedure: Standard surgery

INTERVENTIONS:
Behavioral: Pre-operative use of virtual reality headset — Patient use the virtual reality headset the day before and / or the day of the surgery
  Arms: Immersive reality group
Procedure: Standard surgery — Patient are operated as needed for treatment of colorectal cancer (usual care)
Behavioral: Post-operative use of virtual reality headset — Patient use the virtual reality headset as many time as they want after the surgery during a maximum of 30 days
  Arms: Immersive reality group

SUMMARY:
In patients operated for colorectal cancer, pain, anxiety and depression are important factors in postoperative rehabilitation. The use of new technologies, as virtual reality immersion, could further improve their postoperative management. To date, no study has evaluated the potential benefits of using virtual reality before and after colorectal cancer surgery. The main objective is to determine if virtual reality can reduce postoperative anxiety in patients undergoing colorectal cancer surgery.

To answer this question, the investigators plan to execute a randomized controlled, single-center, open-label, superiority interventional trial. Patients will be randomized into 2 parallel arms: 1 interventional "virtual immersion" arm and 1 "control" arm.

Patients with colorectal cancer, regardless of oncological stage, or a colorectal lesion deemed endoscopically unresectable, with an indication for elective surgical management by laparotomy or laparoscopy will be included.

For patients in the interventional arm, virtual reality headset is put on the day before the operation and in the morning just before going down to the operating theatre. Colorectal cancer surgery then proceeds as usual. In the postoperative period, virtual reality sessions are offered every day and on request without any limit in number. Virtual reality immersion offers a visual and auditory experience during a soothing journey through visual worlds filmed in natural environments. This is a purely contemplative mode, lasting maximum 30 minutes.

For the control arm, patients are treated according to the usual practices of the department and do not have access to virtual reality.

The main purpose is to show a greater decrease in anxiety in the interventional group by measuring the absolute difference between the State-Trait Anxiety Inventory scores before surgery and at discharge.

DETAILED DESCRIPTION:
The investigators plan to execute a randomized controlled, single-center, open-label, superiority interventional trial. Patients will be randomized into 2 parallel arms: 1 interventional "virtual immersion" arm and 1 "control" arm.

Randomization (1:1) will be stratified by cancer type (colon vs rectum). The randomization list will be balanced by small blocks of different sizes, randomly alternated to make it unpredictable. The block sizes will be provided in the final study report. The randomization list will be created by a member of the Digestive and Oncological Surgery department not involved in the study and will be added in REDCap software.

Study process:

- Preoperative consultation: information, surgery planning, obtaining patient consent, randomization and provision of 2 self-administered questionnaires: State-Trait Anxiety Inventory (STAI A "state" anxiety - French version) and CES-D (Center for Epidemiologic Studies - Depression - French version) to be completed at home.

Note: measures of depression (CES-D, Center for Epidemiologic Studies - Depression - French version) and alcohol and tobacco consumption are included. These are indeed confounding factors of anxiety and potential moderating factors of virtual reality's effectiveness.

* Beginning of the study (7 days before surgery): all patients filled in the self-questionnaires at home and brought them the day of the surgery.
* For the interventional arm, patients receive care according to the usual practices of the department as well as virtual reality. Virtual reality immersion offers a visual and auditory experience during a soothing journey through visual worlds filmed in natural environments. Virtual reality headset is put on the day before the operation and in the morning just before going to the operating theatre (only on the morning of the operation for patients hospitalized the same day). The colorectal cancer surgery then proceeds as usual. In the postoperative period, virtual reality sessions are offered every day and on request without any limit in number (day and night). Virtual reality sessions take place in the patient's room in bed or in the armchair on a fixed point, with a maximum duration of 30 minutes. The patient can stop the session at any time. The masks are cleaned before and after each use (Anios® wipes) and brought to the patient by the medical or paramedical staff (nurses only). Virtual reality sessions are prescribed by the medical staff using the software used in the department (Dxcare®). For each session, nurses record the duration of the session, the level of anxiety before the session (numerical scale with a score between 0 and 10), the reasons for a potential refusal, the tolerance and any comments on the programs used.
* For the control arm: patients are treated according to usual practices of the department and do not have access to virtual reality.
* End of study: at the end of the hospitalization, the patients fill in the same self-questionnaire State-Trait Anxiety Inventory (STAI A anxiety "state" - French version). In case of prolonged hospitalization for any reason, the end date of study, with the completion of the questionnaire, is set to the 30th postoperative day.
* No specific post-interventional follow-up is required for this research. The patients included in this study will continue their usual follow-up according to their initial condition and the department's procedures.

The main purpose is to show a greater decrease in anxiety in the interventional group by measuring the absolute difference between the State-Trait Anxiety Inventory scores before surgery and at discharge.

Sample size calculation:

* Control group: decrease of 2.55 points (STAI after-STAI before).
* Intervention group: decrease of 3.1875 points (STAI after-STAI before).
* With a relative difference of 25% (i.e. a difference of 0.6375 +/- 1.2) between the two groups, for an alpha risk of 5% and a power of 80%, 57 patients per arm are required, i.e. a total of 114 patients. To overcome the missing data risk, a 10% addition of patients was estimated, i.e. 124 patients in total.

The main analysis will be an intention-to-treat and per-protocol method. The primary endpoint will be compared between groups by linear regression adjusted for stratification factor and the STAI score at D-7. The application conditions will be checked by studying the residuals. No interim analysis is planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal cancer (colon or rectum), regardless of oncological stage and neo-adjuvant treatments received, or a colorectal lesion judged as endoscopically unresectable, with indication for surgical management either by laparotomy or laparoscopy
* Elective surgery
* Patient ≥ 18 years old
* Patient affiliated to a social security system or entitled to it
* Patient who has received full information on the research organization and has given written consent

Exclusion Criteria:

* Complicated tumour (perforation, occlusion) requiring emergency surgery
* Non-French speaking patient
* Patient subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* Pregnant or breastfeeding woman
* Patient benefiting from the AME
* Epilepsy
* Severe visual or hearing impairment that does not allow the use of headphones
* Autism spectrum disorder
* Claustrophobia
* Confusion
* Medical history of schizophrenia, schizotypal disorders and delusional disorders, and/or patients requiring treatment with : Neuroleptics (Abilify = Aripiprazole and Abilify Now, Clopixol = Zuclopenthixol, Haldol = Haloperidol and Haldol Decanoas, Largactil = Chlorpromazine, Leponex = Clozapine, Loxapac = Loxapine, Nozinan = Levomepromazine, Risperdal = Risperidone and Xeplion and Trevicta, Solian = Amisulpride, Tercian = Cyamemazine, Tiapridal = Tiapride, Xeroquel = Quetiapine, Zyprexa = Olanzapine and Zypadhera); Thymoregulators (Depakote / Depamide = Valproate de Sodium, Lamictal = Lamotrigine, Tegretol = Carbamazepine, Teralithe = Lithium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Anxiety assessment | Up to 30 days
  Change from State-Trait Anxiety Inventory (STAI-A) scores at D-7 before surgery and at discharge (maximum at day 30 after surgery).

SECONDARY OUTCOMES:
Total painkiller use (opioids and non-opioids) during hospitalization | Up to 30 days
  painkillers and their use are prescribed and referenced in the software used in our department (Dxcare®). Data will be collected every day to obtain daily and total consumption.
Pain assessment | Up to 30 days
  Maximum pain experienced by the patient during the hospital stay using the numerical pain scale (NPS): nurses record patients' pain at least 4 times a day and note it directly in Dxcare® software (NPS 0 = no pain, NPS 10 = maximal pain) .
Total anxiolytic use (benzodiazepines, related hypnotics, hydroxyzine) during hospitalization | Up to 30 days
  Anxiolytics and their use are prescribed and referenced in the software used in our department (Dxcare®). Data will be collected every day to obtain daily and total consumption.
Adverse effects of virtual reality immersion | Up to 30 days
  Main adverse effects expected (nausea, vomiting, vertigo, headaches). Virtual reality sessions will be subject to a medical prescription on the software used in our department (Dxcare®). To validate each session, nurses will have to answer a questionnaire stating session duration, anxiety level before the session, reasons for a potential refusal, tolerance, possible comments on the programs used and number of sessions per day.
Morbidity and mortality | Up to 30 days
  Severe morbidity (Clavien Dindo classification)
Confounding factors of anxiety | 7 days before surgery
  Measures of depression (CES-D, Center for Epidemiologic Studies - Depression - French version) and alcohol and tobacco consumption are included. These are indeed confounding factors of anxiety and potential moderating factors of virtual reality's effectiveness.
Morbidity | Up to 30 days
  Transit recovery time

CONTACTS AND LOCATIONS:
Overall Officials: Gilles MANCEAU, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital européen Georges-Pompidou AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Mols F, Schoormans D, de Hingh I, Oerlemans S, Husson O. Symptoms of anxiety and depression among colorectal cancer survivors from the population-based, longitudinal PROFILES Registry: Prevalence, predictors, and impact on quality of life. Cancer. 2018 Jun 15;124(12):2621-2628. doi: 10.1002/cncr.31369. Epub 2018 Apr 6. PMID 29624635
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] Bradt J, Dileo C, Myers-Coffman K, Biondo J. Music interventions for improving psychological and physical outcomes in people with cancer. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD006911. doi: 10.1002/14651858.CD006911.pub4. PMID 34637527
- [Background] Parker S, Zipursky J, Ma H, Baumblatt GL, Siegel CA. A Web-based Multimedia Program Before Colonoscopy Increased Knowledge and Decreased Anxiety, Sedation Requirement, and Procedure Time. J Clin Gastroenterol. 2018 Jul;52(6):519-523. doi: 10.1097/MCG.0000000000000958. PMID 29095417